CLINICAL TRIAL: NCT00002380
Title: A Phase I/II Pharmacokinetic and Safety Study of Saquinavir Soft Gelatin Capsules and Pediatric Pellet Formulations in Combination With Nucleoside Antiretroviral Agents With or Without Nelfinavir, in HIV-Infected Infants and Children
Brief Title: The Safety and Effectiveness of Two Forms of Saquinavir Combined With Other Anti-HIV Drugs in HIV-Infected Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 229K; NV 15445
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Dosage Forms; Saquinavir; Nelfinavir; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; Saquinavir

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Saquinavir

SUMMARY:
To determine the pharmacokinetic properties, tolerance and safety of 2 formulations of saquinavir, given in combination with 2 nucleoside antiretroviral drugs (part 1) or in combination with nelfinavir and nucleoside antiretroviral drugs (part 2), in HIV-infected infants and children.

DETAILED DESCRIPTION:
This Phase I/II study will be conducted in 2 parts each lasting at least 24 weeks. Pharmacokinetics and safety data for part 1, a treatment regimen containing saquinavir and nucleoside antiretrovirals, will be collected for 8 weeks before proceeding to part 2. During the first 8 weeks, pharmacokinetic data will be analyzed to allow dose adjustments for individual patients and to confirm the starting dose estimates for part 2. In addition, safety data will be reviewed to ensure that saquinavir is well tolerated with nucleoside antiretrovirals before it is combined with a second protease inhibitor. In part 2, saquinavir will be combined with nelfinavir, a protease inhibitor recently approved for use in children. The pharmacokinetics and safety profile of these drugs in combination will be determined.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection according to standard definitions employed by the Pediatric AIDS Clinical Trials Group.
* Laboratory evidence of immunosuppression (Centers for Disease Control and Prevention [CDC] categories 2 and 3), or symptomatic HIV disease (CDC categories A, B, and C).
* At least 4 patients (2 in each parts 1 and 2) will be enrolled in each of three age strata:
* 6 months to 2 years; greater than 2 years to 6 years; and greater than 6 years to 13 years. NOTE:
* For the purposes of analysis only, patients will be stratified by age.

  1. Patients must be protease inhibitor therapy naive.
* Antiretroviral agents other than those prescribed by the investigator.
* Biologic response modifiers (other than erythropoietin, G-CSF, short course [<14 days] corticosteroids, or intravenous immune globulin).
* Other investigational drugs.
* Drugs known to significantly interact with saquinavir and/or nelfinavir. Patients must be protease inhibitor therapy naive.

Ages: 6 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28

CONTACTS AND LOCATIONS:
Locations (1):
- Hoffmann - La Roche Inc, Nutley, New Jersey, United States